CLINICAL TRIAL: NCT03486431
Title: A Phase I Dose-escalation Trial of Stereotactic Ablative Body Radiotherapy (SABR) for Non-spine Bone & Lymph Node Oligometastates
Brief Title: A Dose-escalation Trial of Stereotactic Ablative Body Radiotherapy for Non-spine Bone & Lymph Node Oligometastates
Acronym: Destroy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Research Antwerp (Other)
Responsible Party: Principal Investigator, Piet Dirix, Radiation Oncologist, Cancer Research Antwerp
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTOR17007GZA
Record Dates: First submitted 2018-03-19; First posted 2018-04-03 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Cancer
Keywords: Stereotactic Ablative Body Radiotherapy (SABR)
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: 3+3 phase I trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Level I (Experimental): 5 x 7 Gy SABR
  Interventions: Radiation: Stereotactic Ablative Radiotherapy (SABR)
- Level II (Experimental): 3 x 10 Gy SABR
  Interventions: Radiation: Stereotactic Ablative Radiotherapy (SABR)
- Level III (Experimental): 1 x 20 Gy SABR
  Interventions: Radiation: Stereotactic Ablative Radiotherapy (SABR)

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy (SABR) — A minimum of thirty patients will be included for each dose level. An interval of at least 24 weeks from the first patient treatment to the next patient treatment at each dose level will be respected. In the meantime, more patients will be included in the previous dose level, in an effort to establish the secondary endpoints. In case 1-5 patients present with dose-limiting toxicity (DLT) at 6 months after SABR, thirty additional patients will be included at the same dose level. The maximal tolerated dose will be defined as the dose level below which at least 10 patients present with a dose-limiting toxicity at 6 months after SABR.

SUMMARY:
Stereotactic ablative body radiotherapy (SABR) can be considered for patients with so-called "oligometastatic" disease. However, since this is a relatively new technique, information on the optimal scheduling is lacking. Even prospective randomized trials on SABR for oligometastases typically allow different fractionation schedules to be used. This is especially true for non-spine bone and lymph node metastases, where the literature is scarce to non-existent.

There is also emerging evidence that SABR can stimulate the immune response, by a variety of mechanisms such as increasing TLR4 expression on dendritic cells, increasing priming of T cells in draining lymph nodes, and increasing tumor cell antigen presentation by dendritic cells. Again, it is not clear which fractionation schedule elicits the most robust immune response.

Therefore, it is opportune to compare the most commonly used stereotactic regimens regarding toxicity, efficacy, and immune priming.

This trial is a non-randomized prospective phase I trial determining a regimen of choice for patients with non-spine bone and lymph node oligometastases (≤ 3 lesions). The metastatic lesion(s) must be visible on CT and < 5 cm in largest diameter. A total of ninety patients will be consecutively included in three different fractionation regimens. They will be offered stereotactic ablative radiotherapy to all metastatic lesions in 5, 3 or 1 fractions. Dose-limiting toxicity (DLT), defined as any acute grade 3 or 4 toxicity, will be recorded as the primary endpoint. Overall acute and late toxicity, quality of life, local control, and progression-free survival are secondary endpoints.

Liquid biopsies will be collected throughout the course of this trial, i.e. at simulation, after each fraction and at 6 months after the end of the radiotherapy. Translational research will focus on assessment of circulating cytokines and flow cytometry analysis of immune cells.

DETAILED DESCRIPTION:
* Background & rationale

Stereotactic ablative body radiotherapy (SABR) is indicated in patients with oligometastatic, oligoprogressive, or traditionally radioresistant disease, who often present with minimal or no associated symptoms [1, 2]. However, since this is a relatively new technique, information on the optimal scheduling is lacking. Even prospective randomized trials on SABR for oligometastatic disease typically allow different fractionation schedules to be used [3]. This is especially true for non-spine bone and lymph node metastases, where the literature is scarce to non-existent and many different schedules are used, even within a single center [4,5].

There is also emerging evidence that SABR can stimulate the immune response, by a variety of mechanisms such as increasing toll-like receptor 4 (TLR4) expression on dendritic cells, increasing priming of T cells in draining lymph nodes, and increasing tumor cell antigen presentation by dendritic cells [6]. Again, it is not clear which fractionation schedule elicits the most robust immune response. For instance, in combination with cytotoxic T-lymphocyte-associated antigen 4 (anti-CTLA-4) immunotherapy, different radiation regimens in two carcinoma models growing in syngeneic mice were compared [7]. Marked differences in induction of tumor-specific T cells and of an abscopal effect were observed. Each regimen had similar ability to inhibit the growth of the irradiated tumor when radiation was used alone. The addition of anti-CTLA-4, however, caused complete regression of the majority of irradiated tumors and an abscopal effect in mice receiving a hypofractionated regimen (3 fractions of 8 Gy) but not in mice treated with a single dose of 20 Gy. An additional fractionated regimen (5 fractions of 6 Gy) was tested, which showed intermediate results. This indicates that a specific therapeutic window may exist for the optimal use of radiotherapy as an immune adjuvant.

It seems an opportune moment to compare the most commonly used stereotactic regimens regarding toxicity and efficacy.

- Trial design

A minimum of thirty patients will be included for each dose level. An interval of at least 24 weeks from the first patient treatment to the next patient treatment at each dose level will be respected. In the meantime, more patients will be included in the previous dose level, in an effort to establish the secondary endpoints. In case 1-5 patients present with dose-limiting toxicity (DLT) at 6 months after SABR, thirty additional patients will be included at the same dose level. The maximal tolerated dose will be defined as the dose level below which at least 10 patients present with a dose-limiting toxicity at 6 months after SABR.

* Trial procedures

Registration of toxicity: Pre-study; last day of SABR; 3 months after SABR; 6 months after SABR; every 3 months (first year after SABR); every 6 months (second year after SABR); yearly thereafter.

Registration of QoL: Pre-study; last day of SABR; 3 months after SABR; 6 months after SABR; every 3 months (first year after SABR); every 6 months (second year after SABR); yearly thereafter.

Blood sample: every SABR fraction; 3 months after SABR; 6 months after SABR Imaging: 6 months after SABR. All imaging is considered standard and should minimally include a CT of the irradiated lesion(s) but might also include MRI and/or PET-CT (with whatever relevant tracer) if standard for that malignancy.

- Translational research

At the moment, much is unknown about the mechanism of radiotherapy and of SABR in particular. Moreover, only a few predictive biomarkers of response to radiotherapy have been suitably investigated in clinical settings and none of these biomarkers is currently employed in the clinic to assist patient, dose or schedule selection. Hence, liquid biopsies will be collected throughout the course of this study for biobanking.

An interesting measure of DNA damage in circulating tumor cells (CTCs) is γ-H2AX, a biomarker for radiation-induced DNA double-strand breaks [9]. It is also becoming clear that - besides mediating cytotoxic and cytostatic effects on malignant cells - radiotherapy has multipronged immunomodulatory functions manifesting locally (within irradiated lesions) and systemically (within non-irradiated lesions and in the circulation). However, the mechanisms by which radiation induces anti-tumour T cells remain unclear. Apparently, DNA exonuclease Trex1 is induced by radiation doses above 12-18 Gy in different cancer cells, and attenuates their immunogenicity by degrading DNA that accumulates in the cytosol upon radiation. Cytosolic DNA stimulates secretion of interferon-b by cancer cells following activation of the DNA sensor cGAS and its downstream effector STING. Repeated irradiation at doses that do not induce Trex1 amplifies interferon-b production, resulting in recruitment and activation of Batf3-dependent dendritic cells [10]. This effect is essential for priming of CD8+ T cells that mediate systemic tumour rejection (abscopal effect). These data suggest a link between the immune-stimulatory effects of radiation and the DNA damage response.

1. Required samples

   The liquid biopsy in this study encompasses pheripheral blood samples (1x 9mL EDTA and 1x 9mL CPT tubes), to be taken at at simulation, immediately after each fraction, approximately 48 hours after the last fraction, and at 3 and 6 months follow-up for biobanking.
2. Assessment of circulating cytokines

   One EDTA blood tube generally yields 4 mL of plasma, which can be split in half for circulating free DNA (cfDNA) analysis (vide infra) and for the measurement of protein concentrations of circulating cytokines. This latter can be done using Luminex assays, and requires and input volume of 100 µL per assay, allowing 20 cytokines to be profiled using 2 mL of plasma. The plasma must be kept at -80° C. Under these conditions, most cytokines are stable for up to two years under the premises that freeze-thaw cycles are avoided [11].
3. cfDNA for shallow whole genome sequencing

   For cfDNA low-pass whole genome sequencing, cfDNA first needs to be extracted from plasma samples with a typical starting volume of 1 mL. The cfDNA concentrations from 1mL of plasma, in a final elution volume of 50 µL, are highly variable and depend on tumour burden (range 0.2ng/µL to 62.8ng/µL). Hence the calculated cfDNA yield from 1 mL of plasma ranges from 10 ng to 3,140 ng. For low-pass whole genome sequencing using the Thru-PLEX DNA-seq Library Kit, 2 ng of cfDNA is required, suggesting that 1 mL of plasma should be sufficient in most cases. To avoid patient drop-out due to insufficient starting material, biobanking 2 mL of plasma aliquoted in units of 400 µL at -80oC is advisable. An exemplary analysis is provided in Li et al, Mol Oncology, 2017 [12].
4. Flow cytometry analysis of immune cells

   Peripheral blood mononuclear cells (PBMC) can be isolated from heparinized venous blood by centrifugation on a Ficoll-Hypaque gradient within 4 h of venepuncture. The PBMCs can cryopreserved in liquid nitrogen in heat-inactivated foetal bovine serum (FBS) supplemented with 10% dimethyl sulphoxide (DMSO) until analysis. Upon analysis, cells are thawed by submersion at 37° for 1-2 minutes and resuspended in a medium containing Iscove's Modified Dulbecco's Medium (IMDM) supplemented with 20% FBS and 1% glutamine [13].

   - Ethics & regulatory approval

   The trial will be conducted in compliance with the principles of the Declaration of Helsinki (64th WMA General Assembly, Fortaleza, Brazil, October 2013), the principles of GCP and all of the applicable regulatory requirements. The study protocol will be amended to the Ethics Committee (EC) of the GZA Hospitals, Belgium. Any subsequent protocol amendment will be submitted to the EC for approval.

   - Data handling

   All data will be prospectively collected by the clinical trials oncology (www.clinicaltrialsoncology.be) of the GZA hospitals, campus Sint Augustinus.

   - Publication policy

   Publications will be coordinated by the Principle Investigator (PD) and the co-investigators (PM & DV). Authorship to publications will be determined in accordance with the requirements published by the International Committee of Medical Journal Editors and in accordance with the requirements of the respective medical journal.

   - Insurance/Indemnity

   In accordance with the Belgian Law relating to experiments on human persons dated May 7, 2004, Sponsor shall assume, even without fault, the responsibility of any damages incurred by a Study Patient and linked directly or indirectly to the participation to the Study, and shall provide compensation therefore through its insurance.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old with histologically confirmed malignancy.
* Patients with radiosensitive malignancy (e.g. breast, prostate,…) and oligometastases (i.e. ≤ 3 metastases) OR patients with radioresistant malignancy (e.g. renal cell carcinoma, melanoma,…) and an unlimited number of metastases.
* Metastatic lesion must be visible on CT and < 5 cm in largest diameter.
* Patients with ECOG performance status ≤ 1.
* Patients who have received the information sheet and signed the informed consent form.
* Patients must be willing to comply with scheduled visits, treatment plan, and other study procedures.
* Patients with a public health insurance coverage.

Exclusion Criteria:

* Patients with life expectancy < 6 months.
* Patients with previous radiotherapy to the metastatic area excluding stereotactic re-irradiation to the required dose level.
* Patients with significantly altered mental status or with psychological, familial, sociological or geographical condition potential hampering compliance with the study.
* Individual deprived of liberty or placed under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Dose-limiting Toxicity | 6 months after SABR
  To determine the maximum tolerated dose (MTD). The maximal tolerated dose will be defined as the dose level below which at least 10 patients present with a dose-limiting toxicity .

SECONDARY OUTCOMES:
Acute toxicities following SABR | at 3 and 6 months after last day of SABR
  Acute toxicity will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Late toxicities following SABR | at 9, 12, 18 and 24months after last day of SABR
  Late toxicity will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Local control | at 6 months after last day of SABR
  Local response will be evaluated by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. Local failure will be scored as an event if an irradiated lesion shows an increase in size of ≥20%, according to RECIST v1.1.
Progression-free survival | at 6 months after last day of SABR
  Progression-free survival is defined as the time from inclusion to documented disease progression according to RECISTv1.1 or any other clinically relevant definition (e.g. biochemical progression in prostate cancer) or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Piet Dirix, MD, Principal Investigator — Cancer Research Antwerp
Locations (1):
- GZA St Augustinus, Wilrijk, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will allow trial-related monitoring, audits, EC review, and regulatory inspections (where appropriate) by providing direct access to source data and other documents (i.e. patients' case sheets, blood test reports, X-ray reports, histology reports etc.). The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Corbin KS, Hellman S, Weichselbaum RR. Extracranial oligometastases: a subset of metastases curable with stereotactic radiotherapy. J Clin Oncol. 2013 Apr 10;31(11):1384-90. doi: 10.1200/JCO.2012.45.9651. Epub 2013 Mar 4. No abstract available. PMID 23460715
- [Background] Tree AC, Khoo VS, Eeles RA, Ahmed M, Dearnaley DP, Hawkins MA, Huddart RA, Nutting CM, Ostler PJ, van As NJ. Stereotactic body radiotherapy for oligometastases. Lancet Oncol. 2013 Jan;14(1):e28-37. doi: 10.1016/S1470-2045(12)70510-7. PMID 23276369
- [Background] Palma DA, Haasbeek CJ, Rodrigues GB, Dahele M, Lock M, Yaremko B, Olson R, Liu M, Panarotto J, Griffioen GH, Gaede S, Slotman B, Senan S. Stereotactic ablative radiotherapy for comprehensive treatment of oligometastatic tumors (SABR-COMET): study protocol for a randomized phase II trial. BMC Cancer. 2012 Jul 23;12:305. doi: 10.1186/1471-2407-12-305. PMID 22823994
- [Background] Alongi F, Arcangeli S, Filippi AR, Ricardi U, Scorsetti M. Review and uses of stereotactic body radiation therapy for oligometastases. Oncologist. 2012;17(8):1100-7. doi: 10.1634/theoncologist.2012-0092. Epub 2012 Jun 20. PMID 22723509
- [Background] Owen D, Laack NN, Mayo CS, Garces YI, Park SS, Bauer HJ, Nelson K, Miller RW, Brown PD, Olivier KR. Outcomes and toxicities of stereotactic body radiation therapy for non-spine bone oligometastases. Pract Radiat Oncol. 2014 Mar-Apr;4(2):e143-e149. doi: 10.1016/j.prro.2013.05.006. Epub 2013 Jun 29. PMID 24890360
- [Background] de la Cruz-Merino L, Illescas-Vacas A, Grueso-Lopez A, Barco-Sanchez A, Miguez-Sanchez C; Cancer Immunotherapies Spanish Group (GETICA). Radiation for Awakening the Dormant Immune System, a Promising Challenge to be Explored. Front Immunol. 2014 Mar 14;5:102. doi: 10.3389/fimmu.2014.00102. eCollection 2014. PMID 24672524
- [Background] Dewan MZ, Galloway AE, Kawashima N, Dewyngaert JK, Babb JS, Formenti SC, Demaria S. Fractionated but not single-dose radiotherapy induces an immune-mediated abscopal effect when combined with anti-CTLA-4 antibody. Clin Cancer Res. 2009 Sep 1;15(17):5379-88. doi: 10.1158/1078-0432.CCR-09-0265. Epub 2009 Aug 25. PMID 19706802
- [Background] Benedict SH, Yenice KM, Followill D, Galvin JM, Hinson W, Kavanagh B, Keall P, Lovelock M, Meeks S, Papiez L, Purdie T, Sadagopan R, Schell MC, Salter B, Schlesinger DJ, Shiu AS, Solberg T, Song DY, Stieber V, Timmerman R, Tome WA, Verellen D, Wang L, Yin FF. Stereotactic body radiation therapy: the report of AAPM Task Group 101. Med Phys. 2010 Aug;37(8):4078-101. doi: 10.1118/1.3438081. PMID 20879569
- [Background] Martin OA, Anderson RL, Russell PA, Cox RA, Ivashkevich A, Swierczak A, Doherty JP, Jacobs DH, Smith J, Siva S, Daly PE, Ball DL, Martin RF, MacManus MP. Mobilization of viable tumor cells into the circulation during radiation therapy. Int J Radiat Oncol Biol Phys. 2014 Feb 1;88(2):395-403. doi: 10.1016/j.ijrobp.2013.10.033. Epub 2013 Dec 5. PMID 24315565
- [Background] Vanpouille-Box C, Alard A, Aryankalayil MJ, Sarfraz Y, Diamond JM, Schneider RJ, Inghirami G, Coleman CN, Formenti SC, Demaria S. DNA exonuclease Trex1 regulates radiotherapy-induced tumour immunogenicity. Nat Commun. 2017 Jun 9;8:15618. doi: 10.1038/ncomms15618. PMID 28598415
- [Background] de Jager W, Bourcier K, Rijkers GT, Prakken BJ, Seyfert-Margolis V. Prerequisites for cytokine measurements in clinical trials with multiplex immunoassays. BMC Immunol. 2009 Sep 28;10:52. doi: 10.1186/1471-2172-10-52. PMID 19785746
- [Background] Li J, Dittmar RL, Xia S, Zhang H, Du M, Huang CC, Druliner BR, Boardman L, Wang L. Cell-free DNA copy number variations in plasma from colorectal cancer patients. Mol Oncol. 2017 Aug;11(8):1099-1111. doi: 10.1002/1878-0261.12077. Epub 2017 Jun 6. PMID 28504856
- [Background] Chevolet I, Speeckaert R, Schreuer M, Neyns B, Krysko O, Bachert C, Van Gele M, van Geel N, Brochez L. Clinical significance of plasmacytoid dendritic cells and myeloid-derived suppressor cells in melanoma. J Transl Med. 2015 Jan 16;13:9. doi: 10.1186/s12967-014-0376-x. PMID 25592374
- [Derived] Mercier C, Claessens M, Buys MSc A, Gryshkevych S, Billiet C, Joye I, Van Laere S, Vermeulen P, Meijnders P, Lofman F, Poortmans P, Dirix L, Verellen D, Dirix P. Stereotactic Ablative Radiation Therapy to All Lesions in Patients With Oligometastatic Cancers: A Phase 1 Dose-Escalation Trial. Int J Radiat Oncol Biol Phys. 2021 Apr 1;109(5):1195-1205. doi: 10.1016/j.ijrobp.2020.11.066. Epub 2020 Dec 8. PMID 33307151
- [Derived] Mercier C, Dirix P, Meijnders P, Vermeulen P, Van Laere S, Debois H, Huget P, Verellen D. A phase I dose-escalation trial of stereotactic ablative body radiotherapy for non-spine bone and lymph node metastases (DESTROY-trial). Radiat Oncol. 2018 Aug 20;13(1):152. doi: 10.1186/s13014-018-1096-9. PMID 30126440